CLINICAL TRIAL: NCT06639295
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase III Clinical Study to Evaluate the Efficacy and Safety of 611 in Patients With Chronic Rhinosinusitis With Nasal Polyps (CRSwNP)
Brief Title: A Study to Evaluate 611 in Patients With Chronic Rhinosinusitis With Nasal Polyps
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSGJ-611-CRS-III-01
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Sinusitis; Nasal Polyps
MeSH Terms: conditions — Sinusitis; Nasal Polyps | interventions — entacapone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 611 (Experimental): 611 2ml Q2W, subcutaneous (SC) injection
  Interventions: Drug: 611
- Placebo (Placebo Comparator): Placebo subcutaneous (SC) injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 611 — 611 subcutaneous (SC) injection.
  Arms: 611
Drug: Placebo — Placebo subcutaneous (SC) injection.
  Arms: Placebo

SUMMARY:
This study will evaluate the effect and safety of 611 in patients with Chronic Rhinosinusitis with Nasal Polyps (CRSwNP)

DETAILED DESCRIPTION:
The main purpose is to evaluate the effect of 611 on a background of mometasone furoate nasal spray (MFNS) in reducing endoscopic nasal polyp score (NPS) and nasal congestion/obstruction score (NCS) severity in eligible patients with CRSwNP whose disease remains inadequately controlled despite daily treatment with intranasal corticosteroid (INCS) therapy in comparison to placebo

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients aged ≥18 and ≤ 75 years at the time of screening.
* Bilateral CRSwNP.
* Bilateral NPS of ≥5 with a minimum score of 2 in each nasal cavity
* Nasal Congestion Score of 2 at screening and a weekly average severity of 2 at time of randomization.
* Patients whose bilateral sino-nasal polyposis remains inadequately controlled despite prior treatment with SCS anytime within the past 2 years; and/or had a medical contraindication/intolerance to SCS; and/or received nasal polyp surgery 6 months before signing the ICF.

Exclusion Criteria:

* Patients with other nasal diseases or symptoms.
* Patients who are taking or have taken the following prohibited therapies as specified, e.g., systemic steroids within 4 weeks prior to screening, less than 3 months or 5 half-lives for biologic therapy prior to screening.
* Patients who have active Hepatitis B, Hepatitis C or HIV infections as determined by positive results at Screening.
* History of cancer.
* Known or suspected history of immunosuppression.
* Known with allergic or intolerant to mometasone furoate spray or 611/ placebo

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline at Week 24 in Bilateral Nasal Polyp Score (NPS) | 24 weeks
  NPS is evaluated by nasal endoscopy. For each nostril, NPS is graded based on polyp size from 0 = no polyps to 4 = large polyps causing complete obstruction of inferior nasal cavity; lower score = smaller sized polyps. Bilateral NPS is the sum of right and left nostril scores, ranges from 0 (no polyps) to 8 (large polyps), higher score = more severe disease
Change From Baseline at Week 24 in Nasal Congestion Symptom Severity Score (NCS) | 24 weeks
  NCS is assessed by the participants daily from visit 1 and throughout the study on a scale of 0 to 3, where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms, with higher scores indicates more severity.

SECONDARY OUTCOMES:
Change From Baseline to the End of study in Lund Mackay Score | through study completion, an average of 13 months
  The Lund Mackay Score scoring system rates each of both the left and right frontal, maxillary, sphenoid, ostiomeatal complex, anterior ethmoid and posterior ethmoid sinuses using following grading: 0 = normal, 1 = partial opacification, 2 = total opacification. The total score is the sum of scores from each side and ranges from 0 (normal) to 24 (more opacified); higher score indicated more severe disease
Change From Baseline to the End of study in Total Nasal Symptom Score (TNSS) | through study completion, an average of 13 months
  TNSS is a composite of nasal congestion, loss of smell, and rhinorrhea (anterior/posterior nasal discharge), each access on 0-3 categorical scale (where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms). Total score ranges from 0 (no symptoms) to 12 (severe symptoms). Higher score indicated more severe symptoms.
Change From Baseline to the End of study in the University of Pennsylvania Smell Identification Test (UPSIT) Score | through study completion, an average of 13 months
  The UPSIT is a 40-item test to measure the individual's ability to detect odors. Total score ranges from 0 (anosmia) to 40 (normal sense of smell), lower score indicated severe smell loss
Change From Baseline to the End of study in 22-item Sino-nasal Outcome Test (SNOT-22) Scores | through study completion, an average of 13 months
  The SNOT-22 is a validated questionnaire that used to assess the impact of chronic rhinosinusitis phenotype with nasal polyps (CRSwNP) on health-related quality of life (HRQoL). It is a 22 item questionnaire with each item assigned a score ranging from 0 (no problem) to 5 (problem as bad as it can be). The total score may range from 0 (no disease) to 110 (worst disease), lower scores representing better health related quality of life
Adverse events (AEs), measurement of vital signs，physical examination，electrocardiogram and laboratory tests at each visit. | through study completion, an average of 13 months
  The incidence and severity of treatment emergent adverse event (TEAE), including Serious Adverse Event (SAE), as well as clinical symptoms, and any abnormalities of vital signs, physical examinations，electrocardiogram，laboratory tests and, etc.
611 Concentration in Serum | through study completion, an average of 13 months
  The concentration of 611 in Serum

CONTACTS AND LOCATIONS:
Locations (1):
- Site 01, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No